CLINICAL TRIAL: NCT03442764
Title: A Randomized, Double-blind, Placebo-controlled, Concentration-guided, Exploratory Study of Mavacameten in Patients With Symptomatic Non-Obstructive Hypertrophic Cardiomyopathy (nHCM) and Preserved Left Ventricular Ejection Fraction
Brief Title: A Phase 2 Study of Mavacamten in Adults With Symptomatic Non-Obstructive Hypertrophic Cardiomyopathy (nHCM)
Acronym: MAVERICK-HCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MyoKardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYK-461-006
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Non-obstructive Hypertrophic Cardiomyopathy
MeSH Terms: interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Active Treatment for participants with base target trough concentration
  Interventions: Drug: mavacamten
- Group 2 (Experimental): Active Treatment for participants with higher target trough concentration
  Interventions: Drug: mavacamten
- Placebo (Placebo Comparator): Placebo Group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mavacamten — MYK-461
  Other Names: MYK-461
  Arms: Group 1; Group 2
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, exploratory, randomized, double-blind study of the administration of mavacamten in 60 participants with symptomatic nHCM randomized to receive a 16-week course of mavacamten doses titrated to achieve 1 of 2 target drug concentrations.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with nHCM (hypertrophied and non-dilated left ventricle in absence of systemic or other known cause), with LV wall thickness ≥ 15mm at Screening or ≥ 13mm with a positive family history of HCM.
* Age 18 and greater, Body weight > 45kg
* Documented LVEF ≥ 55% at the Screening as determined by echo central lab
* LVOT gradient < 30 mmHg at rest AND during Valsalva AND post-exercise
* NYHA functional class II or III
* Elevated NT-proBNP at rest

Key Exclusion Criteria:

* History of syncope, sustained ventricular tachyarrhythmia with exercise, obstructive coronary artery disease or myocardial infarction within the past 6 months
* History of resuscitated sudden cardiac arrest at any time or known appropriate implantable cardioverter defibrillator (ICD) discharge within 6 months prior to Screening
* Current treatment with disopyramide or ranolazine (within 14 days prior to Screening)
* Current or planned treatment during the study with a combination of beta-blockers and calcium channel blockers
* Has been treated with invasive septal reduction (surgical myectomy or percutaneous alcohol septal ablation [ASA]) within 6 months prior to Screening
* History of resting or post-exercise LVOT >30 mmHg unless subsequently treated by septal reduction
* Has QTc Fridericia (QTcF) >480 ms or any other ECG abnormality considered by the investigator to pose a risk to participant safety (eg, second-degree atrioventricular block type II)
* Has persistent or permanent atrial fibrillation not on anticoagulation for at least 4 weeks prior to Screening and/or not adequately rate-controlled within 1 year of Screening
* History of clinically significant malignant disease within 10 years such as non-metastatic cutaneous squamous cell or basal cell carcinoma
* History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the investigator or MyoKardia physician, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myokardia Medical Information Team, Study Director — MyoKardia, Inc.
Locations (32):
- United States (32):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center (Smidt Heart Institute), Los Angeles, California
  - Stanford Hospital and Clinics/Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Northwestern University, Evanston, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - University of Iowa Hospitals and clinics, Iowa City, Iowa
  - University of Maryland Medical System, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Winthrop Hospital, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Cardiology at Southpoint, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's Cardiology Associates, Bethlehem, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor St. Luke Medical Center at Houston, Texas Heart Institute Out-patient Clinic, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Unity Point Health Meriter Heart and Vascular Institute, Madison, Wisconsin

REFERENCES:
- [Derived] Ho CY, Mealiffe ME, Bach RG, Bhattacharya M, Choudhury L, Edelberg JM, Hegde SM, Jacoby D, Lakdawala NK, Lester SJ, Ma Y, Marian AJ, Nagueh SF, Owens A, Rader F, Saberi S, Sehnert AJ, Sherrid MV, Solomon SD, Wang A, Wever-Pinzon O, Wong TC, Heitner SB. Evaluation of Mavacamten in Symptomatic Patients With Nonobstructive Hypertrophic Cardiomyopathy. J Am Coll Cardiol. 2020 Jun 2;75(21):2649-2660. doi: 10.1016/j.jacc.2020.03.064. PMID 32466879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 157 participants were assessed for eligibility and 59 were enrolled from 35 sites in the United States.
Pre-assignment Details: 59 participants were randomized and 58 entered the treatment period.
Groups:
- Group 1: Received active 16-week course of mavacamten doses titrated to achieve target drug concentrations of ~200 ng/ml. Dose adjustments were done at Week 6 based on PK
- Group 2: Received active 16-week course of mavacamten doses titrated to achieve target drug concentrations of ~500 ng/ml. Dose adjustments were done at Week 6 based on PK
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Placebo
Started | 19 | 21 | 19
Completed | 18 | 21 | 19
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.7) | 50.0 (14.7) | 53.8 (18.2) | 53.9 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 13 | 34
  Male | 10 | 9 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 5
  Not Hispanic or Latino | 18 | 19 | 15 | 52
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 17 | 18 | 17 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 4
NT-proBNP [Mean (Standard Deviation); unit: ng/L] | 1160.7 (859.02) | 933.3 (719.41) | 1164.1 (817.70) | 1080.8 (791.97)
Troponin-I [Number; unit: participants]
  Elevated | 6 | 7 | 6 | 19
  Detectable Not Elevated | 6 | 10 | 5 | 21
  Undetectable | 6 | 4 | 8 | 18
  Missing | 1 | 0 | 0 | 1
New York Heart Association (NYHA) Functional Classification [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) functional classification (class I, II, III or IV) is an established grading scale that classifies patients according to the severity of their symptoms during physical activity. The NYHA functional classification clinically worsens with class increments (more physical activity limitation due to symptoms) and clinically improves with class reductions (less physical limitation due to symptoms). At baseline, all subjects were NYHA Class II or III.
  Participants
    Class II | 15 | 18 | 13 | 46
    Class III | 4 | 3 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment Emergent Adverse Event (TEAE)
Description: This is the percentage of participants who experienced at least one treatment emergent adverse event (TEAE)
Time Frame: From first dose to 8 weeks following last dose (Up to 24 weeks)
Population: All treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Placebo
Number analyzed (Participants) | 18 | 21 | 19
percentage of participants | 88.9 | 90.5 | 68.4

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Serious Treatment-emergent Adverse Event (STEAE)
Description: This is the percentage of participants who experienced at least one serious treatment-emergent adverse event (STEAE)
Time Frame: From first dose to 8 weeks following last dose (Up to 24 weeks)
Population: All treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Placebo
Number analyzed (Participants) | 18 | 21 | 19
percentage of participants | 11.1 | 9.5 | 21.1

ADVERSE EVENTS:
Time Frame: From first dose to 8 weeks following last dose (Up to 24 weeks)
Groups:
- Group 1 Mavacamten: Received active 16-week course of mavacamten doses titrated to achieve target drug concentrations of ~200 ng/ml (Group 1). Dose adjustments were done at Week 6 based on PK
- Group 2 Mavacamten: Received active 16-week course of mavacamten doses titrated to achieve target drug concentrations of ~500 ng/ml (Group 2). Dose adjustments were done at Week 6 based on PK
- Combined MAVA Treatment Group (Group 1+ Group 2): Received active 16-week course of mavacamten doses titrated to achieve target drug concentrations of ~200 ng/ml (Group 1) or ~500 ng/ml (Group 2). Dose adjustments were done at Week 6 based on PK
Arm/Group | Group 1 Mavacamten | Group 2 Mavacamten | Combined MAVA Treatment Group (Group 1+ Group 2) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21 | 0/39 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/18 | 2/21 | 4/39 | 4/19
Other Adverse Events (participants affected / at risk) | 16/18 | 18/21 | 34/39 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Mavacamten (N=18) | Group 2 Mavacamten (N=21) | Combined MAVA Treatment Group (Group 1+ Group 2) (N=39) | Placebo (N=19)
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2 | 1
Systolic dysfunction (Cardiac disorders) | 0 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 Mavacamten (N=18) | Group 2 Mavacamten (N=21) | Combined MAVA Treatment Group (Group 1+ Group 2) (N=39) | Placebo (N=19)
Palpitations (Cardiac disorders) | 1 | 5 | 6 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1 | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 5 | 3
Seasonal Allergy (Immune system disorders) | 1 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 4 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 2
Tooth abscess (Infections and infestations) | 2 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 4 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tooth Fracture (Infections and infestations) | 1 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0
Blood pressure abnormal (Investigations) | 1 | 0 | 1 | 0
Blood urea increased (Investigations) | 1 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Carotid artery dissection (Nervous system disorders) | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 4 | 7 | 1
Head Discomfort (Nervous system disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 1 | 0
Stress (Psychiatric disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 3
Hyperactive pharyngeal reflex (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT03442764/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT03442764/SAP_001.pdf